CLINICAL TRIAL: NCT07254091
Title: Pilot Study of an Implantable Microdevice for In Situ Evaluation of Drug Response in Patients With Pancreatic Cancer
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-0695
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Pharmaceutical Preparations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): This is a single institution pilot study to be performed on a limited number of patients (10) to establish safety and feasibility. There will be only one cohort of patients included and one intervention, the insertion of the microdevice prior to resection of the specimen with the device implanted. All patients will receive this intervention, thereby eliminating any potential bias on confounders.
  Interventions: Combination Product: Device Arm with Therapeutic Agents

INTERVENTIONS:
Combination Product: Device Arm with Therapeutic Agents — Devices manufactured by the Jonas Lab containing microdoses (1/100,000th standard dosage) of chemotherapy agents will be implanted and remain in situ for 4 hours, after which resection of the tumor and corresponding microdevice(s) are removed. The chemotherapeutic agents include Doxorubicin, Gemcitabine , Paclitaxel, 5 Fluorouracil , Oxaliplatin, and Irinotecan.

SUMMARY:
Predicting drug response offers an opportunity to improve cancer treatment delivery. Recently, microdevices were invented to ascertain in vivo drug response but have not yet been evaluated for pancreatic cancer. This study is a prospective phase 1 safety study of intraoperative placement and retrieval of a microdevice in patients with pancreatic cancer. The devices will be implanted intra-operatively and removed en-bloc with the tumor after a 4- hour incubation period. Patients will be monitored to ensure that the placement and retrieval of these devices does not increase complication rates within one month of surgery. To assess feasibility, the tissue surrounding the microdevices is then analyzed to determine the diffusion of drugs from the device(s) to surrounding tissue, and whether the chemotherapeutic effect of diffusing chemotherapy drug has an impact on the surrounding tissue. In an exploratory analysis, material from the patient's tumors will be grown into organoids and drug response correlation from organoids will be compared to the response observed from the microdevices.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least or greater than18 years old
* All sexes, genders, races, and ethnic groups are eligible for this trial
* Patients with a suspicious or histologically confirmed pancreatic lesion for which surgery is indicated for either diagnostic or therapeutic purposes, as determined by the treating surgeon
* Patients must be a candidate for pancreatoduodenectomy or pancreatectomy
* Patients must be evaluated by the operating Surgical Oncologist to determine the feasibility of microdevice implantation based on clinical history, extent, and anatomical location of the tumor seen on baseline imaging
* The effects of the microdevice on the developing human fetus is unknown. For this reason and because the therapeutic agents used in this trial are known to be teratogenic, women of childbearing age must agree to have a negative serum pregnancy test within 48 hours prior to operation.
* Patient must be willing and able to understand and sign informed consent for both the surgical resection as well as the proposed research study obtained prior to any procedures
* Males and females of childbearing potential must agree to use effective contraception starting prior to the first day of treatment and continuing for 30 days after the implantation of the microdevice. Additionally, due to the unknown but potential risks of nursing infants secondary to the treatment of the mother with the chemotherapeutic agents used in this study, breastfeeding should be discontinued for a total of 14 days after the insertion of the microdevice.

Exclusion Criteria:

* Patients with a tumor in a location not amenable to placement of the device prior to the removal of the tumor specimen as determined by the Surgical Oncologist
* Any patient that is pregnant at the time of enrollment or operative intervention is excluded due to the known teratogenicity of the medications involved.
* Patients with a history of prior or concurrent second primary malignancy whose natural history or treatment has the potential to interfere with the safety or primary endpoint efficacy assessment of the pancreas cancer
* Patients with metastatic or locally advanced disease on baseline imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety of micro dosing devices placement and retrieval based on adverse events by assessment of adverse events as defined in the CTCAE v5.0. | 1 year
  Safety will be defined by assessment of adverse events as defined in the CTCAE v5.0.
  Any device resulting in:
  * any listed Serious adverse events as defined in section 8.3.2, or
  * two or more grade 3-4 adverse events directly associated with the device or its placement as defined in section 8.3.3.2

SECONDARY OUTCOMES:
1. To determine the feasibility of microdevice analysis after the intra-operative placement and retrieval of the devices with sufficient associated tissue for histopathologic assessment of drug sensitivity. | 1 year
  To determine the feasibility of microdevice placement and retrieval based on the ability to retrieve the device with sufficient tissue, of sufficient quality , for downstream histopathology analysis and interpretation of at least 50% of the device reservoirs

IPD SHARING:
Plan to Share IPD: Undecided